CLINICAL TRIAL: NCT00157001
Title: Feasibility Study of Photopheresis Post Angioplasty
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Atlantic Health System (Other)
Collaborators: Therakos (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R98-09-013
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Stable Angina Pectoris; Unstable Angina Pectoris; Silent Ischemia
MeSH Terms: conditions — Angina, Stable; Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Photopheresis Post Angioplasty

SUMMARY:
The primary objective of the study is to evaluate the difference in 6-month restenosis rates in coronary artery lesions treated by photopheresis in addition to angioplasty with stent placement, as opposed to no photopheresis after angioplasty and stent placement. Restenosis means the closing up again, or narrowing in diameter, of the previously treated artery, which may cause reduced blood flow and the re-occurrence of symptoms. Photopheresis is a therapeutic technique in which a portion of your white blood cells is collected by a blood separation device and exposed to ultraviolet A light, in combination with the drug 8-MOP (8-methoxypsoralen), then returned to you.

The secondary objectives are:

1. To compare the incidence of major adverse cardiac events (MACE) between the three treatment groups for 6 months post-angioplasty. MACE events include death (cardiac related), myocardial infarction, coronary artery bypass graft surgery, repeat angioplasty to the target vessel, hospitalization and clinical symptoms.
2. To evaluate the safety of the treatment by comparing the incidence of acute and subacute thrombosis, bleeding and vascular complications and other non-MACE events every 2 weeks for 6 months post-angioplasty between the three treatment groups.

DETAILED DESCRIPTION:
Atherosclerosis is a condition of the coronary arteries characterized by abnormal lipid and fibrous tissue accumulation in the vessel wall. This pathologic condition may lead to stenosis of the artery. Percutaneous transluminal coronary angioplasty (PTCA) is a standard method of myocardial revascularization in patients with occlusive coronary artery disease.

Restenosis remains one of the main factors determining the long term success of angioplasty. The literature still reports a 35% restenosis rate after single vessel angioplasty.l,2,3 This study will investigate the feasibility of photopheresis therapy as an adjunct to PTCA plus stent placement as a means to reduce the rate of restenosis.

The UVAX® XTS™ Photopheresis System is currently marketed for use in the palliative treatment of the skin manifestations of cutaneous T-cell lymphoma (CTCL) in persons who have not been responsive to other forms of treatment. For this feasibility study, the XTS System will treat extracorporeally circulating leukocyte-enriched blood with ultraviolet light-A (UVA) in the presence of the photoactive drug UVADEX®.

The UVAR XTS Photopheresis System is used to separate the patient's blood into white blood cells, red blood cells and plasma. The red blood cells are returned to the patient. A dose of two hundred micrograms of UVADEX is added to the photoactivating bag. A portion of the plasma and the white blood cells are exposed to UVA light which causes the methoxsalen in the nucleated white blood cells to form covalent bonds in the pyrimidine bases of the DNA, preventing further replication of the cell. After exposure to UVA light, the white blood cells and plasma are returned to the patient Animal and clinical studies suggest that there is an immune response initiated by the reinitiation of the treated white blood cells. The mechanism of the immune response is not clear. It appears that when the lethally injured white blood cells are reinfused into the patient, surface antigens on the abnormal cells cause the host immune system to recognize the clones of the untreated malignant cells. This may result in a true biologic response modification and induction of a favorable immune response to the underlying malignancy.4 The results of clinical studies of CTCL patients treated with a similar procedure show a prolonged clinical remission.

Photopheresis has been shown to affect diseases mediated by an aberrance in the immune system, e.g., scleroderma, HIV infection and CTCL. These diseases involve a variety of serologic abnormalities and cellular and humoral immune dysfunction. For instance, CTCL demonstrates an abnormally elevated CD4 count; scleroderma reveals a decrease in peripheral T cells but an increase in T cells in tissue; and HIV exhibits a falling CD4

percentage. Several of these diseases have been shown to have antibodies against self to DNA and cellular components.5 Atherosclerosis has recently been shown to have as a constituent factor an underlying immune mechanism.6 There exists a close functional relationship between macrophages and T lymphocytes. In fact, lymphocytes have been demonstrated within the plaques of atherosclerotic vessels.7'8 These lymphocytes have been shown to be activated locally, presumably by antigens presented in the context of class II MHC. Such activated T cells may, in turn, modulate the pathogenesis of restenosis post angioplasty.6 Cyclosporin A, a drug which specifically inhibits T cell activation, has been administered in an animal model and has resulted in significant reduction in intimal lesions post angioplasty.9 This may be a reflection of inhibition of T cell activation which results in an inhibition of monocyte/macrophage activation and therefore inhibition of intimal T cell proliferation. Recent evidence suggests that UVA Photochemotherapy may represent a novel approach to control of smooth muscle cell proliferation without producing cytolysis.10,11 Photopheresis has been postulated to specifically down regulate activated clones to T cells.

All prior clinical studies related to cardiovascular treatment conducted to date have shown that photopheresis with UVADEX is a safe treatment modality without serious side effects. Photopheresis has been studied--for the prevention and treatment of acute rejection in heart transplant recipients.12 As a result of treatment, patients experienced a reduction in the number and severity of rejection episodes. Photopheresis therapy also allowed the reduction of daily immunosuppressive therapy. No major side effects were observed. In another study, the use of monthly photopheresis as an adjunct to standard drug therapy following cardiac transplant found a significant decrease in coronary artery intimal thickness at up to two years of follow-up.13 Photopheresis was determined to be safe, well tolerated and did not increase the morbidity in immunosuppressed patients.

A previous study of the benefits of photopheresis following PTCA enrolled 62 patients (29 treated with photopheresis and oral methoxypsoralen and 33 control). At 6 months follow-up, the patient group treated with photopheresis exhibited fewer clinical signs of restenosis. No significant side effects were observed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a single or multiple de novo coronary artery lesion with 70% stenosis intended to be treated by PTCA using balloons, laser or atherectomy devices plus stent insertion.
* Patients with stable angina pectoris or unstable angina pectoris
* Patients must have veins with adequate access for photopheresis.

-Patients must not be pregnant Female patients who are in child- bearing years and have not been surgically sterilized will be tested for pregnancy by a serum HCG test prior to enrollment into the study and must agree to practice contraception during her participation in the study.

* Patients must be willing to return for evaluation every two weeks and for all photopheresis treatments if in Groups 2, 3.
* Patients must sign an informed consent form prior to entry into the study.
* Patients must live within commuting distance of the treatment center.
* Patients must not be treated with any other investigational drug or device within 6 months prior to participation in this study.

Angiographic Inclusion Criteria:

-Patients who have a single or multiple de novo coronary artery lesion with 70% stenosis successfully treated by PTCA plus stent insertion to <50% stenosis as documented by on-line quantitative coronary angiography (QCA).

General Exclusion Criteria:

* Patients who cannot tolerate extracorporeal volume loss during the leukocyte enrichment phase.
* Patients with photosensitive disease, such as porphyria or systemic lupus erythematous. Care must be taken in selecting patients who require drugs either topically or systemically during the course of the study with photosensitizing potential, such as phenothiazine, tetracycline, sulfonamides or chlorothiazide. Patients who must take photosensitizing drugs will not receive them prior to each photopheresis treatment.
* Patients with renal insufficiency (creatinine >3.0 mg/dl).
* Patients who are pregnant or nursing a child.
* Patients with a severe coexisting medical, physiological or sociological condition that in the opinion of the investigators would preclude any of the procedures contained in this protocol.
* Patients who exhibit idiosyncratic or hypersensitivity reactions to psoralen compounds.
* Patients with a platelet count < 50,000/mm.
* Patients with active hepatitis.
* Patients with hemoglobin < 9 or hematocrit <27.
* Patients under age 18.
* Patients with ostial lesions.
* Patients who are insulin-dependent diabetics.
* Patients who have had an acute myocardial infarction within the previous 8 weeks. is (CCS Class 1, 2, or 4 and Braunwald Class 1-3, B-C) or document silent ischemia.
* Patents must have evidence of left ventricular ejection fraction of >30%.
* Patients must have a hematocrit >27 and hemoglobin >9.
* Patients must be at least 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2000-08; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the difference in 6-month restenosis rates in the treatment of at least a single or multiple de novo coronary artery lesion by photopheresis as an adjunct to angioplasty plus stent insertion in comparison

SECONDARY OUTCOMES:
The primary endpoint will be the six month composite incidence of death from any cause: nonfatal myocardial infarction, ischemia documented by treadmill exercise testing with or w/o nuclear myocardial imaging, or the need for a repeat revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Emil Bisaccia, MD, Principal Investigator — Morristown Memorial Hospital-Atlantic Health System
Locations (1):
- Morristown Memorial Hospital, Morristown, New Jersey, United States